CLINICAL TRIAL: NCT02130154
Title: Brown Adipose Tissue Activity Young and Older Individuals
Brief Title: Brown Adipose Tissue Activity and Age
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, F Holleman, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL 42422.018.12 METC 2012.319
Record Dates: First submitted 2014-03-20; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Obesity; Ageing
Keywords: Brown adipose Tissue; Ageing; Sympathetic Nervous Stimulation; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Young males: Healthy, Lean, Caucasian, Young males
  Interventions: Other: 18-FDG PET CT scan and 123I-MIBG SPECT scan
- Old males: Healthy, Lean, Caucasian, Older males
  Interventions: Other: 18-FDG PET CT scan and 123I-MIBG SPECT scan

INTERVENTIONS:
Other: 18-FDG PET CT scan and 123I-MIBG SPECT scan

SUMMARY:
In this study the investigators aim to investigate whether the sympathetic stimulation of BAT, as assessed with a 123I-metaiodobenzylguanidine single-photon emission computed tomography computed tomography scan, differs between young and elderly subjects, as an explanation for the diminished metabolic brown adipose tissue activity in the elderly.

The investigators hypothesis is that sympathetic nervous system activity in the elderly is diminished as compared to their younger counterparts as an explanation for the diminished metabolic brown adipose tissue activity in the elderly.

DETAILED DESCRIPTION:
The sympathetic nervous system is the primary activator of Brown Adipose Tissue.

Elderly are known to have less metabolically active brown adipose tissue as compared to their younger counterparts.

The reason for this diminished metabolic brown adipose tissue activity is unknown.

However, a lower sympathetic nervous system activation to brown adipose tissue in the elderly might explain a diminished metabolic brown adipose tissue.

Therefore, in this study, both the sympathetic nervous system activation to brown adipose tissue and the metabolic activity will be measured in young and older subjects.

sympathetic nervous system activity will be measured using 123I-metaiodobenzylguanidine single-photon emission computed tomography computed tomography scans, metabolic activity will be measured using 18F- fluorodeoxyglucose positron emission tomography CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Caucasian origin
* Subjects should be able and willing to give informed consent
* 18-65 years old
* BMI range of 19-27 kg/m2

Exclusion Criteria:

* Renal failure (creatinine>135mmol/l)
* Daily use of prescription medication
* Prior participation in a research protocol involving radiation exposure in the last 2 years

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Caucasian Males
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Difference in sympathetic stimulation to BAT between young and older individuals | Participants will be followed for a mean duration of 2 weeks (the maximal time period between the two scans) The outcome measurements will be assessed when the last subject has been scanned approximately one year after starting the trial.

SECONDARY OUTCOMES:
Difference in correlation between sympathetic stimulation of BAT as assessed with 123I-MIBG SPECT scans and metabolic BAT activity as assessed with 18F-Fluorodeoxyglucose(FDG)- positron emission tomography(PET)-CT scan in young and older individuals | Participants will be followed for a mean duration of 2 weeks (the maximal time period between the two scans) The outcome measurements will be assessed when the last subject has been scanned approximately one year after starting the trial.
  The difference in correlation between sympathetic stimulation of BAT as assessed with a MIBG SPECT-CT scan, and BAT activity itself as assessed with 18F-FDG-PET-CT, between young and elderly subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands